CLINICAL TRIAL: NCT06750744
Title: Predictors of Antimicrobial Resistance in the Respiratory Intensive Care Unit of Alexandria Main University Hospital
Status: Completed | Type: Observational
Sponsor: Mohamed Sabry (Other)
Responsible Party: Sponsor-Investigator, Mohamed Sabry, Lecturer of chest diseases, Alexandria University
Organization: Alexandria University (Other)
Other Study IDs: AMR-AMUH
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Identify the Predictors of Antibiotic Resistance
MeSH Terms: interventions — X-Rays; Microbial Sensitivity Tests; Tigecycline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- only one group of patients: to identify the predictors of antibiotic resistance using rates of resistance,comprehensive data of each patient chest X ray,CT,ultrasound
  Interventions: Radiation: chest x ray; Drug: Tigecycline (Tygacil)

INTERVENTIONS:
Radiation: chest x ray — chest X ray identify severity of pneumonia
  Other Names: antibiogram
Radiation: chest X ray — chest radiological evaluation via x ray
Drug: Tigecycline (Tygacil) — selective antibiogram

SUMMARY:
The goal of this clinical trial is to identify the predictors of antibiotic resistance whether clinical or laboratory or radiological or all

DETAILED DESCRIPTION:
The goal of this clinical trial is to identify the predictors of antibiotic resistance like the history of previous antibiotic ,the antibiogram of the centre , comorbidities,..etc to decide the suitable antibiotic

ELIGIBILITY:
Inclusion Criteria:

* Adult patient admitted to the respiratory ICU due to bacterial infection.

  * Recent antibiotic intake in the past three months.
  * Intercostal tube insertion for empyema.
  * Shocked patients with inserted central venous catheter.
  * Intubated or tracheostomized patients.
  * Patients with grade two to four bed sores.

Exclusion Criteria:

* . Inability to provide written informed consent for the study.

  * Non sterile sample collection technique.
  * Inability to provide antibiogram.
  * Isolated patients due to suspected tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The current study aims to identify the predictors of antibiotic resistance in the respiratory intensive care unit of Alexandria main university hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
antibiogram | 3 months
  resistance rates in antibiograms

OTHER OUTCOMES:
resistance rates in the antibiogram | 3 months
  culture and different antibiotic senstivity

CONTACTS AND LOCATIONS:
Overall Officials: mohamed sabry eltarhony, lecturer, Principal Investigator — Alexandria University
Locations (1):
- Chest Department -Faculty of Medicine, Alexandria, Azarita, Egypt

IPD SHARING:
Plan to Share IPD: No
because the facility, where i do my work, refuse to share any project untill it is fully published

REFERENCES:
- See also: antimicrobial resistancde prediction — https://pubmed.ncbi.nlm.nih.gov/17482984/
- Available data/document: Study Protocol: msabry776@yahoo.com — https://pubmed.ncbi.nlm.nih.gov/17482984/ — very good